CLINICAL TRIAL: NCT04039984
Title: Prospective Evaluation of Fixation of the Prime Acetabular Cup
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decided the study on this implant was no longer relevant
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Douglas Naudie, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113456
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Osteoarthritis, Hip
Keywords: radiostereometric analysis; implant migration; total hip replacement; arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: This study design will be a prospective cohort with a retrospective control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prime Cup (Experimental): The study group will receive a Prime cementless acetabular cup (manufactured by Microport located in Arlington, Tennessee). All patients will also receive a cementless Profemur femoral stem with a 32 mm CoCr femoral head, articulating on a highly crosslinked acetabular liner.
  Interventions: Device: Prime Cup

INTERVENTIONS:
Device: Prime Cup — Patients in this group will have the Prime cementless acetabular cup used during surgery.

SUMMARY:
This is a prospective study to compare migration of the Microport Prime acetabular cup to a well-established acetabular cup design after total hip replacement. We will enroll 30 patients with the Prime cup and compare migration, function, pain and quality of life to a historical cohort of patients whom had a different cup used during surgery.

DETAILED DESCRIPTION:
The gold standard for measurement of implant fixation over time is radiostereometric analysis (RSA). At the time of surgery, 0.8-1.0 mm Tantalum beads (typically n = 6-8 per region of interest) are inserted into the bone surrounding the implant of interest, and occasionally also into the polyethylene liner or insert of the implant. RSA exams are then acquired within the first 2 weeks post-operation, and again at 6 weeks, 3 months, 6 months, 1 year, and 2 years. Each exam involves a stereo x-ray acquisition with a calibration unit to reconstruct the 3D location of the implant relative to the marker beads. Across each exam, the migration of the implant relative to the marker beads is tracked compared to the baseline exam acquired within the first 2 weeks. RSA is extremely precise and accurate, and is able to track migrations on the order of 10's of microns. Large early migrations within the first 1-2 years post-operation are predictive of eventual implant loosening and failure. For acetabular cups, proximal migration of greater than 1.0 mm within the first 2 years post-operation is considered unacceptable, with cups migrating between 0.2 and 1.0 mm at risk of having a revision rate exceeding 5% at 10 years.

An RSA study should be completed for any new implant under the principles of phased innovation in orthopaedics. This ensures the new device will achieve long-term, stable fixation prior to its widespread adoption. Many device manufacturers incorporate the results of the RSA migration study into their marketing material. The advantage of RSA is its high degree of accuracy and its well-established thresholds for implant migration, meaning a relatively small number of patients are required to provide meaningful results.

Several joint replacement companies (Microport excluded) have previously released new products to the marketplace without RSA evaluation and these implants have later been identified as having ingrowth problems. The scientific aim of this study is to prove efficacy of ingrowth with a recently released implant.

This study design will be a prospective cohort with a retrospective control group. The study will be conducted at a single centre (London Health Sciences Centre - University Hospital, London, Ontario, Canada) with all cases performed by a single, fellowship-trained high-volume surgeon.

The study group will receive a Prime cementless acetabular cup (manufactured by Microport located in Arlington, Tennessee). All patients will also receive a cementless Profemur femoral stem with a 32 mm Cobalt Chromium femoral head, articulating on a highly crosslinked acetabular liner. The control group will be a previously published cohort that received the Reflection cementless acetabular cup with Roughcoat coating (Smith & Nephew, Memphis, TN). This is a well-established cup with long-term survivorship available in multiple registries, making it an ideal comparator.

Demographic details will be recorded from each patient. Outcome scores will be collected pre-operatively and at each post-operative visit. Standard outcome scores at our centre are the Western and McMaster Universities Osteoarthritis Index (WOMAC), Short Form 12 (SF-12), and Harris Hip Score. At the time of surgery, n = 8 of 1.0 mm Tantalum beads will be inserted into the pelvis surrounding the acetabular cup. Patients will undergo post-operative supine RSA exams within 0-2 weeks (baseline exam) and at 6 weeks, 3 months, 6 months, 1 year, and 2 years, following standardized protocols. RSA exams will be conducted at Robarts with a member of the research team escorting participants over to Robarts for each required post-operative visit.

ELIGIBILITY:
Inclusion Criteria:

* hip osteoarthritis
* scheduled for primary total hip arthroplasty
* ability to provide informed consent
* over the age of 18 years

Exclusion Criteria:

* prior arthroplasty on the indicated joint
* individuals who do not speak or understand English
* individuals with neuromuscular disorders or cognitive impairments
* individuals ho live >100km from our centre and/or are unlikely to return for multiple follow-up appointments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Implant Migration | 2 years
  Migration will include translations, rotations and maximum total point motion measured between the 3D CAD models of the cup and the bone bead segment using model-based RSA software

SECONDARY OUTCOMES:
Short Form 12 | 2 years
  Patient-reported questionnaire to assess general health and quality of life. Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Western Ontario and McMaster Universities Osteoarthritis Index | 2 years
  Patient-reported questionnaire to assess function, stiffness and pain caused by hip or knee osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales (function, stiffness and pain). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The total score is calculated by summing the scores for each subscale. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Harris Hip Score | 2 years
  The Harris Hip Scale (HHS) was developed for the assessment of the results of hip surgery, and is intended to evaluate various hip disabilities and methods of treatment in an adult population. It is a physician-completed instrument that consists of subscales for pain severity (1 item, 0-44 points), function (7 items, 0-47 points), absence of deformity (1 item, 0-4 points), and range of motion (2 items, 0-5 points). The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. The maximum score possible is 100.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Naudie, MD, Principal Investigator — London Health Sciences Centre

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share individual participant data.

REFERENCES:
- [Background] Valstar ER, Gill R, Ryd L, Flivik G, Borlin N, Karrholm J. Guidelines for standardization of radiostereometry (RSA) of implants. Acta Orthop. 2005 Aug;76(4):563-72. doi: 10.1080/17453670510041574. PMID 16195075
- [Background] Pijls BG, Nieuwenhuijse MJ, Fiocco M, Plevier JW, Middeldorp S, Nelissen RG, Valstar ER. Early proximal migration of cups is associated with late revision in THA: a systematic review and meta-analysis of 26 RSA studies and 49 survivalstudies. Acta Orthop. 2012 Dec;83(6):583-91. doi: 10.3109/17453674.2012.745353. Epub 2012 Nov 5. PMID 23126575
- [Background] Malchau H, Bragdon CR, Muratoglu OK. The stepwise introduction of innovation into orthopedic surgery: the next level of dilemmas. J Arthroplasty. 2011 Sep;26(6):825-31. doi: 10.1016/j.arth.2010.08.007. Epub 2010 Oct 2. PMID 20888183
- [Background] Naudie DD, Somerville L, Korczak A, Yuan X, McCalden RW, Holdsworth D, Bourne RB. A randomized trial comparing acetabular component fixation of two porous ingrowth surfaces using RSA. J Arthroplasty. 2013 Sep;28(8 Suppl):48-52. doi: 10.1016/j.arth.2013.06.041. Epub 2013 Aug 13. PMID 23953963